CLINICAL TRIAL: NCT02296112
Title: A Phase II Open-Label, Two-Arm Study of the MEK Inhibitor, Trametinib, to Investigate the Safety and Anti-Cancer Activity in Subjects With Melanoma With BRAF Non-V600 Mutations
Brief Title: Trametinib in Treating Patients With Advanced Melanoma With BRAF Non-V600 Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Douglas Johnson, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC MEL 1457; NCI-2014-02185 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MEL1457; GSK1120212; VICC MEL 1457 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (trametinib) (Experimental): Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: trametinib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; Mekinist
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial studies trametinib in treating patients with melanoma with v-Raf murine sarcoma viral oncogene homolog B (BRAF) non-V600 mutations that has spread to other places in the body. Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical efficacy of trametinib in advanced BRAF nonV600mutation (MUT) melanoma ("high activity" group).

SECONDARY OBJECTIVES:

I. To characterize the safety of trametinib. II. To evaluate the progression-free survival (PFS) and overall survival (OS) of trametinib in advanced BRAF nonV600MUT melanoma.

TERTIARY OBJECTIVES:

I. To determine the clinical efficacy of trametinib in advanced BRAF nonV600MUT melanoma ("low activity/unknown" group).

II. Identify mechanisms of resistance to trametinib in this patient population.

OUTLINE:

Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically or cytologically confirmed diagnosis of melanoma
* BRAF mutation in loci other than V600 (BRAF nonV600 MUT) or BRAF fusion detected by genetic testing of the primary tumor or regional/distant metastasis
* Subjects must provide either a fresh or archived tumor sample for correlative study analyses
* For subjects with melanoma, archived or freshly biopsied tumor tissue (preferred) must be obtained prior to enrollment. Tissue shipment tracking information should be provided before administration of study treatment is initiated. However, if shipping will be delayed and tissue shipment tracking information is unavailable, study drug may be administered prior to tissue receipt pending discussion with principal investigator.
* Measurable disease (i.e., present with at least one measurable lesion per Response Evaluation Criteria In Solid Tumors [RECIST], version 1.1)
* All prior anti-cancer treatment-related toxicities (except alopecia and laboratory values) must be =< grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.0) at the time of randomization. Subjects with endocrinopathies (e.g. hypopituitarism, hypothyroidism, hypoadrenalism) caused by immune therapies currently on adequate hormone replacement WILL be permitted.
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to randomization and agree to use effective contraception
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) > or = 1.0 × 10^9/L
* Hemoglobin > or = 9 g/dL
* Platelet count > or = 75 x 10^9/L
* Prothrombin time (PT)/international normalized ratio (INR)* = or < 1.3 x upper limit of normal (ULN)

  * Subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to randomization; PT and partial thromboplastin time (PTT) > 1.5 x ULN are permitted in these subjects
* PTT =or < 1.3 x ULN
* Albumin >or = 2.5 g/dL
* Total bilirubin = or < 1.5 x ULN
* Alanine aminotransferase (ALT) = or < 2.5 x ULN
* Creatinine = or < 1.5 ULN or calculated creatinine clearance* > or = 50 mL/min

  * Calculate creatinine clearance using standard Cockcroft-Gault formula; creatinine clearance must be > or = 50 mL/min to be eligible
* Left ventricular ejection fraction (LVEF) > or = lower limit of normal (LLN) by echocardiogram (ECHO)

Exclusion Criteria:

* No prior therapy with inhibitors affecting the mitogen-activated protein kinase (MAPK) pathways at any level (BRAF, mitogen-activated protein [MAP]/extracellular signal-related kinase [ERK] kinase [MEK], neuroblastoma RAS viral [v-ras] oncogene homolog [NRAS], ERK inhibitors) for unresectable stage IIIC or stage IV (metastatic) melanoma; no limit to other therapies (immunotherapy or chemotherapy); prior systemic treatment in the adjuvant setting is allowed; (note: ipilimumab treatment must end at least 8 weeks prior to study day 1)
* BRAFV600 mutation positive
* NRAS codon 12, 13, or 61 mutation
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to study day 1, or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to study day 1
* Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to study day 1
* Current use of a prohibited medication as described
* History of another malignancy

  * Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected, non-melanoma skin cancer, or subjects with indolent second malignancies are eligible. T1a melanoma and melanoma in situ are permitted. Consult Medical Monitor if unsure whether second malignancies meet requirements specified above.
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted)
* History of leptomeningeal disease or spinal cord compression secondary to metastasis
* Brain metastasis, unless previously treated with surgery or stereotactic radiosurgery and the disease has been confirmed stable (i.e., no increase in lesion size) for at least 6 weeks with two consecutive magnetic resonance imaging (MRI) scans using contrast prior to study day 1; enzyme inducing anticonvulsants are not allowed while patients are on study treatment
* A history or evidence of cardiovascular risk including any of the following:

  * A QT interval corrected for heart rate using the Bazett's formula (QTc) > or = 480 msec
  * A history or evidence of current clinically significant uncontrolled arrhythmias

    * Exception: subjects with atrial fibrillation controlled for > 30 days prior to study day 1
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study day 1
  * A history or evidence of current >= class I congestive heart failure as defined by the New York Heart Association (NYHA) guidelines
  * Treatment refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy
  * Patients with intra-cardiac defibrillators or permanent pacemakers
  * Known cardiac metastases
* A history or current evidence of retinal vein occlusion (RVO) including:

  * History of RVO or
  * Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO such as:

    * Evidence of new optic disc cupping
    * Evidence of new visual field defects
    * Intraocular pressure > 21 mmHg as measured by tonography
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* History of interstitial lung disease or pneumonitis
* Females who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnson, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (4):
- United States (4):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Nebhan CA, Johnson DB, Sullivan RJ, Amaria RN, Flaherty KT, Sosman JA, Davies MA. Efficacy and Safety of Trametinib in Non-V600 BRAF Mutant Melanoma: A Phase II Study. Oncologist. 2021 Sep;26(9):731-e1498. doi: 10.1002/onco.13795. Epub 2021 May 4. PMID 33861486
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Trametinib)
Started | 9
Completed | 0
Not Completed | 9
Not completed — Disease progression | 7
Not completed — Toxicity | 1
Not completed — Began an alternate therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.111111111111 (5.546381313885)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate in "High Affinity" Group
Description: Per RECIST criteria version (v.) 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions.
Time Frame: Up to 12 months
Population: patients with advanced melanoma with High Activity BRAF Mutations or Fusion Events.
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Groups:
- Treatment (Trametinib) "High Activity": Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  trametinib: Given PO
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
Arm/Group | Treatment (Trametinib) "High Activity"
Number analyzed (Participants) | 2
Proportion of participants | 0.5 [0.026 to 0.974]

2. Secondary Outcome: Progression-Free Survival All Patients
Description: Progression of disease as defined by RECIST 1.1 criteria will be reported. Time from on treatment to progression or death (whichever comes first). For those did not progress or die, they were censored at the last follow up or off study date(if they do not have a last date of follow up).
Time Frame: On-study date to lesser of date of progression or date of death from any cause (assessed up to 3 years)
Population: Patients with advanced melannoma with BRAF non-V600 mutations and received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 9
months | 7.5 [0.99 to NA] — The upper bound for the 95% confidence interval is not estimable from the data.

3. Secondary Outcome: Duration of Response in "High Affinity" Group
Description: Estimated probable duration from date of objective response to date of disease progression, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >= 20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: Date of first partial or complete response as defined by RECIST 1.1 criteria to date of progression up to 3 years
Population: Patients with advanced melanoma with BRAF "high activity"
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib) "High Activity"
Number analyzed (Participants) | 2
months | NA [NA to NA] — Only 1 patient out of 2 had partial response on 6/7/2015. The patient was off study on 12/22/2015 due to alternative therapy and then the status was no longer known.

4. Secondary Outcome: Clinical Benefit (Complete Response [CR] + Partial Response [PR] + Stable Disease [SD]) Per RECIST v. 1.1 in "High Affinity" Group
Description: Per RECIST criteria v. 1.1: measurable lesions: complete response (CR) disappearance of target lesions, partial response (PR) > 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) > 20% increase in the sum of the LD of target lesions or appearance of new lesions, stable disease (SD) neither sufficient decrease nor increase of the sum of smallest sum of the LD of target lesions.
Time Frame: Up to 12 months
Population: patients with advanced melanoma with High Activity BRAF Mutations or Fusion Events.
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment (Trametinib) "High Activity"
Number analyzed (Participants) | 2
Proportion of participants | 0.5 [0.026 to 0.974]

5. Secondary Outcome: Overall Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring.
Time Frame: On-study date to date of death from any cause (assessed up to 3 years)
Population: All patients on study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Trametinib)
Number analyzed (Participants) | 9
months | 27.6 [2.5 to NA] — The upper bound is not estimable from the data.

6. Secondary Outcome: Number of Patients With Each Worst-Grade Toxicity
Description: Safety profile shown by count of patients according to the worst-grade toxicity experienced by each, where worst-grade toxicity is per National Cancer Institute (NCI) common toxicity criteria: grade 1, mild; grade 2, moderate; grade 3, severe; grade 4, life-threatening; grade 5, death.
Time Frame: On-study date to 30 days following final dose of study drug, up to 3 years
Population: All patients on study.
Measure: Number; unit: participants
Groups:
- Treatment (Trametinib) Worst Grade 1: Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  trametinib: Given PO
  laboratory biomarker analysis: Correlative studies
  pharmacological study: Correlative studies
- Worst Grade 2; Worst Grade 3: Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in ...
Arm/Group | Treatment (Trametinib) Worst Grade 1 | Worst Grade 2 | Worst Grade 3
Number analyzed (Participants) | 9 | 9 | 9
participants | 2 | 3 | 3

7. Secondary Outcome: Overall Response Rate in "Low Affinity" Group
Description: as for outcome 4
Time Frame: Up to 12 months
Population: Patients on study with low activity
Measure: Mean (95% Confidence Interval); unit: proportion
Groups:
- Low Activity: Patients with low activity of BRAF mutations
Arm/Group | Low Activity
Number analyzed (Participants) | 7
proportion | 0.14 [0.007 to 0.513]

8. Other Pre Specified Outcome: Duration of Response in "Low Affinity" Group
Description: Estimated probable duration from date of first partial or complete response as defined by RECIST 1.1 criteria to date of disease progression, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >= 20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: Up to 3 years
Population: Patients on study with low activity
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Low Activity
Number analyzed (Participants) | 7
months | NA [NA to NA] — One patient started the treatment on 03/09/2019. Then had partial response. But the date was not known. Then the patient got off the treatment on 05/31/2018 due to toxicity.

9. Other Pre Specified Outcome: Clinical Benefit (CR + PR + SD) Per RECIST v. 1.1 in "Low Affinity" Group
Description: as for outcome 4
Time Frame: Up to 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Molecular Characteristics of Patient Samples, Including Archival Samples
Description: Molecular characterization of tumor tissue will be performed to identify markers that correlate with clinical responsiveness to treatment with trametinib. Optional on-treatment biopsies will be used to evaluate pharmacodynamic and other molecular effects of treatment, which will be compared to clinical outcomes. Optional post-progression samples will be analyzed to identify mechanisms of resistance.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 39 months
Arm/Group | Treatment (Trametinib)
All-Cause Mortality (participants affected / at risk) | 3/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trametinib) (N=9)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Limb edema (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Rash (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trametinib) (N=9)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (11)
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 5 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (20)
Constipation (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Xerosis (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 6 (9)
Feeling cold all the time (General disorders) | 1 (1)
face edema (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Irritability (General disorders) | 1 (2)
Localized edema (General disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 2 (4)
GGT increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
LDH Elevated (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 3 (7)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (3)
Loss of consciousness (for less than a minute during a fall) (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Involuntary movements (Nervous system disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Right shoulder pain (arm pit dull pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Tonsil infection (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Lymphedema (Vascular disorders) | 3 (4)
Hypertension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Shortness of breath (Cardiac disorders) | 1 (1)
Burning sensation on the hands and ears (General disorders) | 1 (1)
Dry skin (General disorders) | 1 (1)
Depression (General disorders) | 1 (1)
Anxiety (General disorders) | 1 (1)
Dyspnea (General disorders) | 1 (1)
Alopecia (General disorders) | 1 (1)
Bloating (General disorders) | 1 (1)
Bloating and gas pain (General disorders) | 1 (1)
Bruising (General disorders) | 1 (1)
Bumps in mouth (General disorders) | 1 (2)
Bumps in nose (General disorders) | 1 (2)
Dry mouth (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Lumbar nerve root injury (General disorders) | 1 (3)
Lymphedema (General disorders) | 1 (1)
Pain in right side chest (Gastrointestinal disorders) | 1 (1)
Platelets elevated (Investigations) | 1 (2)
Total white blood count elevated (Investigations) | 1 (1)
Hyperlipidemia (Investigations) | 1 (1)
Vitamin D deficiency (Investigations) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (3)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (2)
Hypergylcemia (Blood and lymphatic system disorders) | 1 (1)
ALT 402 U/L (Blood and lymphatic system disorders) | 1 (1)
AST 170 U/L (Blood and lymphatic system disorders) | 1 (1)
Toe fungus (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Pain in left upper extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue infection in left arm (Musculoskeletal and connective tissue disorders) | 1 (1)
3rd finger amputation (Musculoskeletal and connective tissue disorders) | 1 (1)
Leg spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Xerostemia (Gastrointestinal disorders) | 1 (1)
New skin lesion (Skin and subcutaneous tissue disorders) | 2 (2)
Toe fungus (Skin and subcutaneous tissue disorders) | 1 (1)
Red elevated papule under the right axilla (Skin and subcutaneous tissue disorders) | 1 (1)
New basal cell carcinoma right flank (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intermittent head pressure (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT02296112/Prot_SAP_000.pdf